CLINICAL TRIAL: NCT01785966
Title: Checklist During Multidisciplinary Daily Visits and Clinician Prompting for Reduction of Mortality in Intensive Care Units: A Cluster Randomized Trial
Brief Title: Checklist During Multidisciplinary Visits for Reduction of Mortality in Intensive Care Units
Acronym: CHECKLIST-ICU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital do Coracao (Other)
Collaborators: Sociedade Hospital Samaritano (Other); D'Or Institute for Research and Education (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 11673812310010060
Record Dates: First submitted 2013-02-01; First posted 2013-02-07 (Estimated); Last update posted 2015-03-04 (Estimated); Status verified 2014-11

CONDITIONS: Critical Care
Keywords: Critical care; quality improvement; checklist

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Daily checklist and clinician prompting (Experimental): Checklist during multidisciplinary daily visits + clinician prompting + audit & feedback
  Interventions: Behavioral: Daily checklist and clinician prompting
- Usual care (No Intervention): Usual care

INTERVENTIONS:
Behavioral: Daily checklist and clinician prompting — Interventions are:
  Checklists: The checklists are arranged in a paper notebook (one per patient) with a daily list on each page, as most ICUs do not have electronic health record systems. During the multidisciplinary visit, the checklist items are read aloud by the nurse and answered by participants of the visit. The checklist is applied at least once on all week days preferably in the mornings, although we strongly suggest applying it also on weekend days.
  Daily Goals and Clinician Prompting: During the clinical discussion of each patient and the application of the checklist, the intensivists write down the daily goals in a standardized form and read them aloud to the team. Every afternoon between 3 and 5 PM, a nurse reviews the daily goals and takes note of any pending items. Subsequently, the nurse prompts the on-call physician, requesting solutions for these pending items.
  Arms: Daily checklist and clinician prompting

SUMMARY:
CHECKLIST-ICU will be a cluster randomized trial to ascertain whether the use of an intervention including 1) checklists with assessment of daily goals during the multidisciplinary visit, and 2) clinician prompting can reduce in-hospital mortality of patients admitted to intensive care units (ICUs).

The investigators also aim to describe participant ICUs in terms of the standards for intensive care units proposed by the Brazilian National Health Agency (ANVISA).

DETAILED DESCRIPTION:
Cluster randomized trial involving ICUs in Brazil. ICU is the unit of randomization.

The trial will have two stages:

* Stage I - Baseline data.In this stage we will:

  * Apply "Safety Attitudes Questionnaire" for the employees of the participating ICU.
  * Characterize participant ICUs in terms of the standards (RDC nº7/2010, RDC nº26/2012 e RDC nº 63/2011) for intensive care units proposed by the Brazilian National Health Agency (ANVISA)
  * Characterize patients: we will collect data from 60 consecutive critically ill patients from each participant ICU to describe adherence to measures aimed at avoiding ICU complications and clinical outcome measures.
* Stage II - Intervention: This is the main stage for data analysis. ICUs will be randomly assigned to an experimental or control group. The experimental group should use a multi-item verbal checklist including assessment of daily goals during the multidisciplinary visits plus clinician prompting. We will collect data from 60 additional patients for each ICU in both study groups and apply "Safety Attitudes Questionnaire".

ELIGIBILITY:
Inclusion criteria for clusters:

* Intensive care units, except dedicated coronary care units/cardiac intensive care units and step-down units;
* Must have multidisciplinary daily rounds or coordinators agree to implement daily rounds, including at least one physician and one nurse, conducted at least on week days.

Exclusion criteria for clusters:

• We will exclude ICUs that systematically apply checklists in the multiprofessional daily visit. We define systematically applied checklist when all the following criteria are met:

* Content: structured evaluation following a digital or printed document of multiple items focused on prevention of common ICU complications (eg. ventilator-associated pneumonia, stress ulcer, venous thromboembolism and/or catheter-associated bloodstream infection) and/or explicit assessment of daily goals;
* Time frame: daily application of checklist for at least 30 days
* Periodicity: at least 3 days per week
* How is applied: verbal, observational (1 professional check all items), with or without written register

Patient inclusion criteria:

• Adult patients (≥18 years-old) with anticipated ICU length of stay > 24 hours.

Patient exclusion criteria;

* High probability of death within 24 hours or patients admitted in ICU for palliative care only;
* Suspected or confirmed brain death.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13637 (Actual)
Dates: Start 2013-08; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
In-hospital mortality truncated at 60 days | Hospital discharge; average of 20 days; follow-up limited to 60 days
  Follow-up will be limited to 60 days after ICU admission. Patients who are still in the hospital after 60 days of ICU admission will be considered as discharged alive.

SECONDARY OUTCOMES:
Head of the bed elevated at 30° | Every 3 three days, from ICU day 2 to 17
Adequate prophylaxis for venous thromboembolism | Every 3 three days, from ICU day 2 to 17
Patient-days under light sedation or alert and calm (RASS - 3 to 0) | Every 3 three days, from ICU day 2 to 17
Rate of central-line catheter use | Daily from ICU day 2 to 17
Indwelling urinary catheter use rate | Daily from ICU day 2 to 17
Rate of patients receiving enteral or parenteral feeding | Every 3 three days, from ICU day 2 to 17
Tidal volume <=8mL/kg of predicted body weight in patients on mechanical | Every 3 three days, from ICU day 2 to 17
ICU mortality | ICU discharge; follow-up limited to 60 days
  Follow-up will be limited to 60 days after ICU admission. Patients who are still in the ICU after 60 days of ICU admission will be considered as discharged alive.
Central line-associated bloodstream infection (CLABSI) rate | Daily from ICU day 2 to 17
  Following the Centers for Disease Control/National Healthcare Safety Network (CDC/NHSN) Surveillance Definition of Healthcare-Associated Infection 2008
Urinary tract infection associated with catheter rate | Daily from ICU day 2 to 17
Ventilator-associated pneumonia (VAP) | Daily from ICU day 2 to 17
Length of ICU stay | Hospital discharge; follow-up limited to 60 days
  Follow-up will be limited to 60 days after ICU admission. Patients who are still in the hospital after 60 days of ICU admission will be considered as discharged alive.
Length of hospital stay | Hospital discharge; average of 20 days; follow-up limited to 60 days
  Follow-up will be limited to 60 days after ICU admission. Patients who are still in the hospital after 60 days of ICU admission will be considered as discharged alive.
Mechanical ventilation-free days at 28 days | Day 28 after ICU admission
  Survival time free of invasive mechanical ventilation from ICU admission to day 28.
  Patients who were discharged from hospital alive before 28 days are considered to be alive and free of mechanical ventilation until the 28th day.
Safety Attitudes Questionnaire Score | In phase 1, between sept/2013 and january/2014 each ICU staff answered the questionnaire once. In phase 2, between july/2014 and december/2014 the questionnaire was applied again (once for each ICU staff).
  Survey

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre B Cavalcanti, MD, PhD, Study Chair — Research Institute - Hospital do Coracao; Fernando Bozza, MD, PhD, Principal Investigator — D'Or Institute for Research and Education; Jorge I Salluh, MD, PhD, Principal Investigator — D'Or Institute for Research and Education; Flávia Machado, MD, PhD, Principal Investigator — Federal University of São Paulo; Edson R Romano, MD, Principal Investigator — Hospital do Coracao; Karina Normilio-Silva, Principal Investigator — Research Institute - Hospital do Coração; Otavio Berwanger, MD, PhD, Principal Investigator — Research Institute - Hospital do Coracao; Patricia Vendramim, R.N., Principal Investigator — Hospital Samaritano; Viviane C Chiattone, RN, Principal Investigator — Research Institute - Hospital do Coracao; Helio P Guimaraes, MD, PhD, Principal Investigator — Research Institute - Hospital do Coracao; Valquiria P Campagnucci, MD, Principal Investigator — Research Institute - Hospital do Coracao; Derek C Angus, MD, PhD, Principal Investigator — Department of Critical Care Medicine and CRISMA Center. University of Pittsburgh School of Medicine; Fernanda Carrara, RN, Principal Investigator — Latin American Sepsis Institute (LASI); Juliana Lubarino, RN, Principal Investigator — Latin American Sepsis Institute (LASI); Aline R Sila, RN, Principal Investigator — D'Or Institute for Research and Education; Grazielle Viana, RN, Principal Investigator — D'Or Institute for Research and Education; Lucas P Damiani, MSc, Principal Investigator — Research Institute - Hospital do Coracao; Chung C Chang, PhD, Principal Investigator — Division of General Internal Medicine at University of Pittsburgh
Locations (1):
- Alexandre Biasi Cavalcanti, São Paulo, São Paulo, Brazil

REFERENCES:
- [Derived] Writing Group for the CHECKLIST-ICU Investigators and the Brazilian Research in Intensive Care Network (BRICNet); Cavalcanti AB, Bozza FA, Machado FR, Salluh JI, Campagnucci VP, Vendramim P, Guimaraes HP, Normilio-Silva K, Damiani LP, Romano E, Carrara F, Lubarino Diniz de Souza J, Silva AR, Ramos GV, Teixeira C, Brandao da Silva N, Chang CC, Angus DC, Berwanger O. Effect of a Quality Improvement Intervention With Daily Round Checklists, Goal Setting, and Clinician Prompting on Mortality of Critically Ill Patients: A Randomized Clinical Trial. JAMA. 2016 Apr 12;315(14):1480-90. doi: 10.1001/jama.2016.3463. PMID 27115264
- [Derived] Damiani LP, Cavalcanti AB, Moreira FR, Machado F, Bozza FA, Salluh JI, Campagnucci VP, Normilio-Silva K, Chiattone VC, Angus DC, Berwanger O, Chou H Chang C. A cluster-randomised trial of a multifaceted quality improvement intervention in Brazilian intensive care units (Checklist-ICU trial): statistical analysis plan. Crit Care Resusc. 2015 Jun;17(2):113-21. PMID 26017129
- [Derived] CHECKLIST-ICU Investigators and BRICNet; Machado F, Bozza F, Ibrain J, Salluh F, Campagnucci VP, Guimaraes HP, Normilio-Silva K, Chiattone VC, Vendramim P, Carrara F, Lubarino J, da Silva AR, Viana G, Damiani LP, Romano E, Teixeira C, da Silva NB, Chang CC, Angus DC, Berwanger O. A cluster randomized trial of a multifaceted quality improvement intervention in Brazilian intensive care units: study protocol. Implement Sci. 2015 Jan 13;10:8. doi: 10.1186/s13012-014-0190-0. PMID 25928627